CLINICAL TRIAL: NCT06268132
Title: Healthy Longevity and Mortality in Long-living Adults: Contributors and Causes - Lifestyle, Socioeconomic Background, and Replicative Aging
Brief Title: Longevity in Russia
Status: Recruiting | Type: Observational
Sponsor: Center for Strategic Planning, of the Federal Medical and Biological Agency (Other)
Collaborators: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MLS90
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: LONGEVITY 1; Frailty; Aging; Age-related Cognitive Decline; Aging Disorder
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, stool, saliva, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-living individuals: Long-living individuals at least 90 years of age from the Central Federal District of Russia

SUMMARY:
This is an observational cohort study of long-living adults (participants aged 90 and above) from the Central Federal District of Russia.

The study seeks to determine the genetic and cellular and molecular determinants of healthy longevity and to assess the impact of lifestyle and socioeconomic and environmental factors on healthy longevity.

The study is expected to result in the development of a panel of markers of healthy longevity and/or a model of healthy aging based on the analysis of all factors under consideration.

DETAILED DESCRIPTION:
The study involves a long-term observation of a cohort of long-living adults. During the first visit, a medical professional will take a detailed medical history and perform a comprehensive geriatric assessment (for 15 geriatric syndromes), and physical examination. The participants will have their biomaterials sampled for basic and extended blood biochemistry testing, telomere length measurement, common urine tests and subsequent biobanking and additional studies: whole genome sequencing, DNA methylation analysis, transcriptome analysis, and 16S RNA sequencing of stool and saliva.

Follow-up checks will be carried out once a year by phone or during additional visits.

The study seeks to identify the genetic, epigenetic, and metagenomic determinants associated with the successful and unsuccessful aging phenotypes, mortality, and survival in long-living individuals.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* 90 years of age or above

Exclusion Criteria:

* Refusal to participate or to provide informed consent;
* Any other criteria deemed reasons for exclusion by the Principal Investigator.

Min Age: 90 Years | Sex: All
Age Groups: Older Adult
Study Population: The inclusion of participants will be carried out with the involvement of social services, boarding houses for labor veterans, geriatric centers and other geriatric services in the central region of Russia
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-12-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality among long-living adults | at least 1 year after inclusion in the study
  Mortality among long-living adults within at least 1 year after inclusion in the study and factors associated with mortality will be assessed.
Morbidity among long-living adults | at least 1 year after inclusion in the study
  Morbidity among long-living adults within at least 1 year after inclusion in the study and factors associated with morbidity will be assessed.

SECONDARY OUTCOMES:
Aging phenotypes | at least 2 years after inclusion in the study
  Identification of successful and unsuccessful aging phenotypes
Social, economic, and medical- history-related determinants | at least 2 years after inclusion in the study
  Identification of social, economic, and medical- history-related determinants of successful and unsuccessful aging, geriatric syndromes
Genetic determinants | at least 2 years after inclusion in the study
  Identification of the genetic determinants of successful and unsuccessful aging, geriatric syndromes
Epigenetic determinants | at least 2 years after inclusion in the study
  Identification of the epigenetic determinants (methylation sites) of successful and unsuccessful aging, geriatric syndromes
Metagenomic determinants | at least 2 years after inclusion in the study
  Identification of the metagenomic determinants (16S-rSeq) of successful and unsuccessful aging, geriatric syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Irina D. Strazhesko, M.D., Ph.D, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- RUSSIAN CLINICAL AND RESEARCH CENTER OF GERONTOLOGY, Pirogov Russian National Research Medical University of the Ministry of Healthcare of the Russian Federation, Moscow, Russia